CLINICAL TRIAL: NCT00862056
Title: Prospective Detection of Subclinical Atherosclerosis in Asymptomatic Individuals With High Likelihood of Coronary Artery Disease With a Novel, Low-Radiation Volumetric Computed Tomography Approach
Brief Title: Detection of Subclinical Atherosclerosis in Asymptomatic Individuals
Acronym: Decide CTA
Status: Completed | Type: Observational
Sponsor: Piedmont Healthcare (Other)
Responsible Party: Sponsor
Other Study IDs: PH08012
Record Dates: First submitted 2009-03-12; First posted 2009-03-16 (Estimated); Last update posted 2017-11-20 (Actual); Status verified 2017-11

CONDITIONS: Coronary Artery Disease
Keywords: asymptomatic; coronary artery disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood for DNA and RNA analysis for genetics and genomics
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cardiac CT: All participants will undergo a coronary artery CT angiogram
  Interventions: Procedure: Cardiac CT

INTERVENTIONS:
Procedure: Cardiac CT — All participants will undergo a coronary artery CT angiogram with contrast.

SUMMARY:
This study will evaluate the use of cardiac CT in identifying atherosclerosis plaque in patients who have not been diagnosed with atherosclerosis and who have no symptoms of the disease but who are at risk of developing atherosclerosis based on traditional risk factors such as diabetes or a family history of coronary artery disease.

ELIGIBILITY:
Inclusion Criteria:

* Males between ages 35-90 or females between ages 40-90
* No known coronary artery disease

  * no prior coronary disease by cardiac catheterization (no more than 40% in any major epicardial vessel)
  * no prior myocardial infarction
  * no prior ST-elevation myocardial infarction (1 mm ST-elevation in 2 contiguous leads)
  * no prior non-ST-elevation myocardial infarction (CK-MB > 2x ULN or elevated troponin that is indicative of myocardial necrosis based on local institutional cutpoints)
  * no prior coronary revascularization procedure
* Aymptomatic

  * no chest pain, shortness of breath, angina or angina-equivalent that is assumed to be related to myocardial ischemia
* Presence of a high-risk feature (at least one of the following four will quality)

  * High FRS ≥20% (http://hp2010.nhlbihin.net/atpiii/calculator.asp)
  * Diabetes Mellitus
  * Premature CAD in a first-degree relative
  * High Risk Lipid Profile (must meet one of the following laboratory criteria)

    1. LDL > 250 mg/dL
    2. HDL < 20 mg/dL
    3. Triglycerides > 1000 mg/dL
    4. LP(a) > 80 mg/dL
* Provide written informed consent and Authorization for Use/Disclosure of PHI

Exclusion Criteria:

* Known genetic form of hypercholesterolemia based on clinical criteria (e.g. familial hypercholesterolemia, etc.)
* Creatinine 1.5 mg/dL or greater
* Irregular rhythm precluding cardiac CT examination
* Uncontrolled hypertension (SBP>210 mmHg or DBP>140 mmHg on treatment)
* Known moderate or severe allergy to iodine-based contrast agents (mild prior reactions that could be treated as an outpatient or that could be prevented by pre-medication in the past do not constitute exclusion)
* Known Pregnancy
* Unwilling or unable to consent
* Presence of any co-morbidity that makes life expectancy less than 24 months
* Unwilling or unable to complete follow-up
* Unwilling or unable to provide written informed consent and Authorization for Use/Disclosure of PHI

Ages: 35 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Coronary Artery Disease
Sampling Method: Non-Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2009-01 (Actual); Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
The primary endpoint of the study is identifying the prevalence of coronary artery disease (CAD) in an asymptomatic population of patients without prior history of, but with high likelihood of CAD. | 6 months, 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Rinehart, MD, Principal Investigator — Piedmont Healthcare
Locations (1):
- Piedmont Hospital, Atlanta, Georgia, United States